CLINICAL TRIAL: NCT06281873
Title: Outpatient Clinic of Alexandria University Teaching Hospital, Egypt
Brief Title: Closure of Oroantral Fistula (OAF) Using Platelet Rich Fibrin With Middle Meatal Antrostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0645
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-03

CONDITIONS: Oroantral Fistula
MeSH Terms: conditions — Oroantral Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- closure of the OAF with PRF application (Experimental): This study was conducted on 9 patients. application of PRF membrane
  Interventions: Procedure: closure by PRF membrane

INTERVENTIONS:
Procedure: closure by PRF membrane — Oral fistulectomy was done with proper curettage. EMMA was performed. closure of the OAF by application of PRF membrane and covering it with an acrylic splint

SUMMARY:
the study evaluated the one stage endoscopic middle meatal antrostomy (EMMA) technique with the application of a platelet rich fibrin membrane (PRF) for Oroantral Fistula (OAF) closure and relief of maxillary sinusitis.

DETAILED DESCRIPTION:
This study was conducted on nine eligible patients who complained of OAF with odontogenic sinusitis. Oral fistulectomy was done with proper curettage. Then, EMMA was performed with simultaneous closure of the OAF by application of PRF membrane and covering it with an acrylic splint. Patients were clinically evaluated for closure of the OAF after 14th days postoperatively, relief of the symptoms, and assessment of the pain level. Also, measurement of the size of the bone defect with the aid of computed tomography (CT) preoperatively and 24th weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1 - Adult patients between the ages of 20-60 years. 2- Patients who were suffering from chronic fistula that occurred after the extraction of upper posterior teeth

Exclusion Criteria:

1. patients who have any systemic disease that contraindicates any intervention under general anesthesia (e.g., coronary artery disease).
2. OAF that occurred as a result of other causes (e.g., cyst,and trauma)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the soft tissue wound's healing | 1st, 7th, and14 days postoperatively
  closure of the fistula using the Clinical Healing Score (CHS). CHS: score ranging from 0-5

SECONDARY OUTCOMES:
Secondary radiographic outcomes, assessment of bone formation | 24 weeks postoperatively
  Measurement of the size of the defect with CT size measured by millimeters (mm)

CONTACTS AND LOCATIONS:
Overall Officials: MONA SAMY, PHD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elgabarty AT, Elmahallawy AS, Ibraheam AA, Oraby MS. Closure of oroantral fistula using platelet rich fibrin with endoscopic middle meatal antrostomy. BMC Oral Health. 2024 Jun 16;24(1):698. doi: 10.1186/s12903-024-04409-0. PMID 38880902